CLINICAL TRIAL: NCT05463965
Title: A Multicenter, Randomized, Double-Blind, Active-Controlled (BOTOX®) and Placebo-Controlled Study to Evaluate the Efficacy and Safety of QM1114-DP for the Treatment of Moderate to Severe Glabellar Lines in Subjects of Chinese Origin
Brief Title: A Study to Evaluate the Efficacy and Safety of QM1114-DP for the Treatment of Moderate to Severe Glabellar Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 43QMCH1908
Record Dates: First submitted 2022-07-14; First posted 2022-07-19 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-04

CONDITIONS: Moderate to Severe Glabellar Lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment Group (Experimental): Single injection with QM1114-DP in glabellar lines
  Interventions: Biological: QM1114-DP
- Active-Controlled Group (Active Comparator): Single injection with BOTOX® in glabellar lines
  Interventions: Biological: OnabotulinumtoxinA
- Placebo-Controlled Group (Placebo Comparator): Single injection with placebo in glabellar lines
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: QM1114-DP — Intramuscular injection
  Arms: Treatment Group
Biological: OnabotulinumtoxinA — Intramuscular injection
  Arms: Active-Controlled Group
Biological: Placebo — Intramuscular injection
  Arms: Placebo-Controlled Group

SUMMARY:
This is a phase 3, multicenter, randomized, double-blind, active-controlled and placebo-controlled study to evaluate the efficacy and safety of 50 units (U) of QM1114-DP for the treatment of moderate to severe GL in male and female subjects of Chinese origin. The study has been designed to test the superiority of QM1114-DP compared to placebo, and the non-inferior efficacy of QM1114-DP compared to onabotulinumtoxinA (BOTOX®), in improving the appearance of moderate to severe GL.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects of Chinese origin from ≥18 to ≤65 years of age.
2. Moderate to severe GL (grade of 2 or 3 on the 4-point Photographic Scale ranging from 0 [none] to 3 [severe]) at maximum frown as assessed by the Investigator (GL-ILA).
3. Moderate to severe GL (grade of 2 or 3 on the Static 4-point Categorical Scale ranging from 0 [no wrinkles] to 3 [severe wrinkles]) at maximum frown as assessed by the subject (GL-SLA).
4. Female of non-childbearing potential (i.e., post-menopausal [absence of menstrual bleeding for 1 year prior to screening, without any other medical reason], or has undergone hysterectomy or bilateral oophorectomy). OR Female of childbearing potential with a negative pregnancy test at screening and baseline, and agrees to use a highly effective and approved contraceptive method for the duration of the study. A highly effective method of contraception is defined as: Bilateral tubal ligation; Combined (estrogen and progesterone containing) oral, intravaginal or transdermal contraceptives that inhibit ovulation as the primary mode of action, on a stable dose for at least 28 days prior to screening visit; Intrauterine device (IUD) inserted at least 28 days prior to screening visit; Intrauterine hormone-releasing system; Partner vasectomized for at least three months prior to screening visit; Progestogen-only oral, injectable or implantable contraceptives that inhibit ovulation as the primary mode of action, on a stable dose for at least 28 days prior to screening visit; or Strict abstinence (i.e., refraining from heterosexual intercourse for the duration of the subject's participation in the study).
5. Time and ability to complete the study and comply with instructions.
6. Understands the study requirements and signed the informed consent form (ICF).

Exclusion Criteria:

1. Previous use of any botulinum neurotoxin (BoNT) in facial areas within 9 months prior to study treatment.
2. Anticipated need for treatment with BoNT of any serotype for any reason during the study (other than the study products).
3. Female who is pregnant, breast feeding, or intends to conceive a child during the study.
4. Known allergy or hypersensitivity to any component of the investigational study products (QM1114-DP or BOTOX®) or any other BoNT serotype.
5. Inability to substantially lessen GL by physically spreading them apart, as determined by the Investigator.
6. Clinically significant abnormal lab finding(s) at screening, or clinically significant abnormal focused physical exam finding(s) at screening or baseline visits, in the opinion of the Investigator.
7. Excessive skin laxity in the treatment area or periorbital area.
8. Previous use of any hyaluronic acid soft tissue augmentation therapy in the glabella or forehead area within 6 months before baseline.
9. Previous soft tissue augmentation with any permanent (non-biodegradable such as silicone, polyacrylamide, etc.) or semi-permanent (i.e., calcium hydroxylapatite, poly-L-Lactic acid or polymethyl-methacrylate) product; lifting threads, or autologous fat in the treatment area.
10. History, presence, or predisposition of eyelid or eyebrow ptosis, amblyopia, or previous surgery around the eye that may lead to the above events, as determined by the Investigator.
11. Marked facial asymmetry, excessive dermatochalasis (i.e., excess of skin in eyelids), or marked periocular or eyebrow asymmetry.
12. Presence of scar(s), piercing(s), or tattoo(s) (including microblading of eyebrow or eyeliner) in the treatment area or around the treatment area that, in the Investigator's opinion, may interfere with study evaluations.
13. Presence of inflammation, active infection or skin disorder such as eczema, rosacea, facial psoriasis, herpes zoster etc., near or in the treatment area.
14. Presence of cancerous or pre-cancerous lesions in the treatment area.
15. History of other facial treatment, surgery or other aesthetic procedures (e.g., ablative skin resurfacing, laser treatment, micro needling, chemical peel) in the previous 12 months that, in the Investigator's opinion, could interfere with study injections and/or assessments.
16. Planned facial surgery, eye surgery (including LASIK procedure) or facial aesthetic procedures (e.g., ablative skin resurfacing, laser treatment, micro needling, chemical peel, BoNT treatment, or dermal fillers) in the face during the study period.
17. History or presence of facial nerve palsy, or any medical condition that may put the subject at increased risk with exposure to BoNT including diagnosed myasthenia gravis, Lambert-Eaton syndrome, amyotrophic lateral sclerosis, or any other condition that might interfere with neuromuscular function.
18. Use of medications that affect neuromuscular transmission such as curare-like depolarizing agents, lincosamides, polymyxins, anticholinesterases, and aminoglycoside antibiotics.
19. Subject with bleeding disorder or subject currently using anticoagulants.
20. Subject has any prior or current psychiatric illness (e.g., Psychosis, depression, anxiety), alcohol or drug abuse, or is taking antidepressant, anxiolytic, or antipsychotic medication that, in the Investigator's opinion, could affect the subject's safety and/or participation in the study.
21. Other concurrent medical conditions, therapy, or other condition that, in the Investigator's opinion, would interfere with the evaluation of the study medication, safety or efficacy, and/or put the subject at risk if he/she participates in the study.
22. Participation in an investigational device or drug study within 30 days prior to study treatment or plans to enroll in any other investigational study during participation in this study.
23. Study site personnel, close relatives of the study site personnel (e.g., parents, children, siblings, or spouse), employees or close relatives of employees at the Sponsor company.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 605 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2023-01-29 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
The composite responder rate will be evaluated at Month 1 using the GL-ILA and the GL-SLA at maximum frown. | 1 month
  A composite responder is defined as a subject who achieves a score of 0 or 1 in GL severity and at least 2 grades improvement from baseline on both the GL-ILA and GLSLA scales concurrently.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wu, Principal Investigator — Peking University First Hospital
Locations (6):
- China (6):
  - Guangdong Second Provincial General Hospital, Guangzhou, Guangdong
  - Xiangya 3rd Hospital, Changsha, Hunan
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Beijing Tongren Hospital, CMU, Beijing
  - Peking University First Hospital, Beijing
  - Tianjin University General Hospital, Tianjin